CLINICAL TRIAL: NCT04678908
Title: A Phase 1, Multicenter, Open-label, Dose-escalation and Dose-expansion Study of the Safety and Pharmacokinetics of HB0025 in Patients With Advanced Solid Tumors
Brief Title: A Study of Injection HB0025 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: HB0025-01
Record Dates: First submitted 2020-12-15; First posted 2020-12-22 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Tumor, Subjects
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HB0025 (Experimental): HB0025 IV every 2 weeks (q2w)
  Interventions: Drug: HB0025

INTERVENTIONS:
Drug: HB0025 — Patients will be assigned to dose regimens in the order of enrollment, and they will receive their assigned fixed dose of HB0025 via intravenous infusion.
  Other Names: Recombinant Humanized Anti-PD-L1 Monoclonal Antibody-VEGFR1 Fusion Protein

SUMMARY:
This is a multicenter, open-label, dose escalation and expansion study. During the study, subjects will be evaluated for safety, toxicity, tolerability, PK/PD, immunogenicity, biomarkers, and antitumor activity of HB0025. The phase I study will enroll up to 154 subjects with advanced solid tumors who have progressed on or after standard of care therapy and for whom there is no further treatment available that in the judgement of the patient's physician would be beneficial. One cycle is defined as 28 days.

DETAILED DESCRIPTION:
Dose escalation phase Approximately 19 to 74 subjects will receive escalating doses on HB0025 monotherapy. The escalating dose phase is composed of an accelerated titration design and a conventional 3+3 design.

During the dose escalation, when a given dose level completes the DLT observation period, an evaluation of PK, PD, biomarkers, tolerability and efficacy will be performed and if this dose level is considered as a possible candidate dose level for OBD. Determination of MTD or OBD will be expanded to a total of 6 subjects (if not already done due to observation of a DLT). After the MTD or OBD is determined, the dose group will continue to recruit subjects until the total number of subjects reaches 10 to confirm that the MTD or OBD is RP2D.

Dose escalation phase Approximately 80 subjects will be enrolled into expansion doses on HB0025. During the dose escalation process, dose expansion studies will be conducted based on the preliminary determination of RP2D and the expanded tumor types.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female. Age ≥ 18 years.
2. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
3. 1) Dose escalation phase: Patients with histologically or cytologically confirmed advanced malignant solid tumor who have received or been intolerant of all standard therapies thought to confer clinical benefit. These solid tumors include but are not limited to hepatocellular carcinoma (HCC), non-small cell lung cancer (NSCLC), renal carcinoma (RCC), endometrial carcinoma, etc.

2) Dose expansion phase:

a) Advanced HCC Cohort:

i) Unresectable HCC with diagnosis confirmed by histology/cytology or clinical criteria.

ii) Assessed by the investigator as likely to benefit from the study drug therapy; and should have progressed at least one prior systemic therapy regimen which could include but not limited to sorafenib, lenvatinib, donafenib, systematic chemotherapy,etc.

iii)Child-Pugh Classification with score ≤ 6 points.(See Appendix13.6 for criteria) VI)HBsAg test is negative.Patients with active hepatitis B virus (HBV) infection must have a viral load < 500 IU/mL within 28 days prior to start of study treatment and be on suppressive therapy (per local standard of care) for a minimum of 14 days prior to start of study treatment and for the length of the study.

b) Advanced Renal Cell Carcinoma Cohort and Advanced Endometrial Carcinoma Cohort:

i) Histopathological and/or cytological diagnosis of patients with advanced clear cell renal carcinoma, advanced endometrial carcinoma, who are not suitable for radical treatment or have relapsed/metastatic disease; Advanced clear cell renal carcinoma should be assessed as medium-high risk by the International Metastatic Renal Cell Carcinoma Database Alliance (IMDC).

ii) Assessed by the investigator as likely to benefit from the study drug therapy Patient with disease progression from at least one previous systemic treatment or who are intolerant to the current standard treatment as determined by the investigator.

c) Other advanced solid tumor cohort: Patient with other advanced solid tumors that are not suitable for radical therapy or relapse /metastasis diagnosed histopathological and/or cytologically according to the type of tumor that responds well during the dose escalation phase.

4. Accelerated escalation: Evaluable disease per RECIST v1.1 for solid tumors; Radiographic disease assessment at baseline can be performed up to 28 days prior to the first dose.

5. 3+3 dose escalation and dose expansion cohort: At least one measurable tumor lesion as per RECIST criteria v1.1 defined as having at least one dimension with a minimum size of 10 mm in the longest diameter by CT or MRI scan for non-nodal lesions or ≥15 mm in short axis for nodal lesions. Radiographic disease assessment at baseline can be performed up to 28 days prior to the first dose.

6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

7. Life expectancy ≥3 months.

8. Adequate hepatic function as evidenced by meeting all the following requirements:

1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN).
2. AST and ALT ≤ 2.5 × ULN; AST or ALT ≤ 5 × ULN if liver metastases are present.

9. Serum creatinine (Scr) < 1.5 × ULN and calculated creatinine clearance (CrCL) > 40 mL/min (Cockroft-Gault Equation).

10. Hematological function defined as:

1. Absolute neutrophil count ≥1,500/µL without growth factor support within 2 weeks prior to the first dose of HB0025.
2. Hemoglobin ≥ 9 g/dL without transfusion or erythropoietin within 2 weeks prior to the first dose of HB0025.
3. Platelet count ≥ 75,000/µL without transfusion or recombinant human thrombopoietin within 2 weeks prior to the first dose of HB0025.

11. Coagulation: International Normalized Ratio (INR)≤1.6 (unless receiving anticoagulation therapy). Subjects on full-dose oral anticoagulation must be on a stable dose (minimum duration 14 days). If receiving warfarin, the subject must have an INR≤3.0 and no active bleeding (ie, no bleeding within 14 days prior to first dose of study drug). Subjects on low molecular weight heparin will be allowed. Subjects must have no active bleeding or clinically significant bleeding within 14 days prior to first dose of study drug.

12. Recovery, to Grade 0-1, from adverse events related to prior anticancer therapy except alopecia, < Grade 2 sensory neuropathy, lymphopenia, and endocrinopathies controlled with hormone replacement therapy.

13. All patients will be required to provide (if available) archived paraffin blocks or at least 10 unstained slides prior to study entry. Patients who do not have available archival tissue will be asked (optional) to provide fresh tissue from core-needle or punch biopsy.

Exclusion Criteria:

Patients who meet any of the following criteria cannot be enrolled:

1. Symptomatic central nervous system metastases; patients with asymptomatic CNS metastases who are radiologically and neurologically stable > 4 weeks following CNS-directed therapy, and are on a stable or decreasing dose of corticosteroids equivalent to < 10 mg prednisone/day for at least 2 weeks prior to study treatment are eligible for study entry.
2. Active autoimmune disease or history of autoimmune disease requiring systemic therapy < 2 years prior to screening except hypothyroidism, vitiligo, Grave's disease, Hashimoto's disease, or Type I diabetes. Patients with childhood asthma or atopy that has not been active in the 2 years prior to study screening are eligible.
3. History of Grade 3-4 immune-related adverse events (irAEs) or irAEs requiring discontinuation of prior therapies, (except for grade 3 endocrinopathy that is managed with hormone replacement therapy).
4. Use of systemic corticosteroids in a dose equivalent to > 10 mg/day of prednisone or other immunosuppressive agent < 2 weeks prior to screening; the use of topical, intraocular, intra-articular, intranasal or inhaled corticosteroids (systemic absorption is low) will be allowed to prevent (e.g., allergy to contrast agents) or treat non-autoimmune condition (e.g. delayed hypersensitivity caused by exposure to allergens).
5. Cerebrovascular accident (CVA), Transient ischemic attack (TIA), myocardial infarction (MI), unstable angina, or New York Heart Association (NYHA) class III or IV heart failure < 6 months of study entry; mean ECG QT-interval corrected according to Fridericia's formula (QTcF) > 470 milliseconds (ms) (males) or > 480 ms (females) obtained from three ECGs; uncontrolled arrhythmia < 3 months of study entry. Patients with rate-controlled arrhythmias may be eligible for study entry at discretion of the Investigator.
6. Uncontrolled diabetes mellitus with hemoglobin A1c > 8%.
7. Subjects who have received previous simultaneous therapy with a PD-1 pathway inhibitor and a macromolecule VEGF inhibitor (Bevacizumab, Ramucirumab, etc).
8. Anticancer therapy or radiation < 5 half-lives or 4 weeks (whichever is shorter) prior to study entry; palliative radiotherapy to a single area < 2 weeks prior to study screening is permitted. Measurable lesions cannot be previously irradiated unless they have demonstrated growth after radiation therapy (RT).
9. Prior stem cell, bone marrow or solid organ transplant.
10. Concurrent malignancy < 5 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, localized prostate cancer, ductal carcinoma in situ of the breast, or < T1 urothelial carcinoma. Patients with prostate cancer that is under active surveillance are eligible.
11. Any of the following infections. 1) Active infection requiring intravenous therapy < 2 weeks prior to screening. 2) Active tuberculosis (via medical history). 3) Positive test for HIV antibody at screening. 4) Active hepatitis B or C. HBV carriers without active disease (HBV DNA titer < 1000 cps/mL or 200 IU/mL), or cured Hepatitis C (negative HCV RNA test) may be enrolled.
12. Major surgery < 4 weeks or minor surgery < 2 weeks prior to screening; wound must be fully healed.
13. History of severe allergic reactions, Grade 3-4 allergic reaction to treatment with another monoclonal antibody, or known to be allergic to protein drugs or recombinant proteins or excipients in HB0025 drug formulation.
14. Live virus vaccines < 30 days prior to screening.
15. Pregnant or breast-feeding females.
16. Any investigational agents or study drugs from a previous clinical study within 30 days of the first dose of study treatment.
17. Any other serious underlying medical condition (e.g. active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders, cardiac conditions), or psychiatric, psychological, familial condition or geographical location that, in the judgment of the Investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.
18. Women of childbearing potential who do not consent to use acceptable methods of birth control during treatment and for an additional 90 days after the last administration of HB0025.
19. Men with a partner of childbearing potential who do not consent to use acceptable methods of birth control during treatment and for an additional 90 days after the last administration of HB0025.

1) Single method i) Intrauterine device (IUD) ii) Vasectomy of a female subject's male partner iii) Contraceptive rod implanted into the skin 2) Combination method (requires use of two of the following) i) Diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide) ii) Cervical cap with spermicide (nulliparous women only) iii) Contraceptive sponge (nulliparous women only) iv) Male condom or female condom (cannot be used together) v) Hormonal contraceptive: oral contraceptive pill (estrogen/progestin pill or progestin -only pill), contraceptive skin patch, vaginal contraceptive ring, or subcutaneous contraceptive injection.

20. Positive COVID-19 qRT-PCR and/or serology test result during screening; 21. Subjects with a history of arterial or deep venous thrombosis within 3 months before enrollment, or patients with evidence or history of bleeding tendency within 2 months before enrollment, regardless of severity.

22. Severe dyspnea or pulmonary dysfunction or need for continuous supportive oxygen inhalation.

23. Skin wound, surgical site, wound site, mucosal ulcer, or fracture not completely healed; 24. Conditions that may cause gastrointestinal bleeding or perforation (such as duodenal ulcer, intestinal obstruction, Crohn's disease, ulcerative colitis, large-scale gastrectomy, etc.); patients with previous history of intestinal perforation and intestinal fistula but not cured after surgical treatment; esophageal and gastric varices.

25. Subjects received immune modulators treatment, including but not limited to cyclosporine and tacrolimus, within 2 weeks before enrollment.

26. Inability to comply with study and follow-up procedures. 27. Patients who have history of interstitial lung disease or non-infectious pneumonitis (except factor of radiation therapy; such patients should be discussed with the Medical Monitor before enrollment.

28. Subjects who in the judgement of the Investigator are not suited to participate in this trial.

29. Uncontrolled arterial hypertension despite standard treatment (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg).

30. Patients with > 2+ protein on urine dipstick should have a 24-hour urine collection; Patients with ≥ 2 g of protein in the urine on 24-hour collection are ineligible for study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-02-02 (Estimated); Study Completion 2024-05-23 (Estimated)

PRIMARY OUTCOMES:
Safety assessment in dose-escalation phase | 240 Days
  Safety profile including adverse events, changes in safety assessment parameters (e.g. incidence of AEs, vital signs, ECGs, clinical laboratory results and DLTs);
Safety assessment in dose-escalation phase | 240 Days
  MTD or OBD and/or RP2D.
Efficacy assessment in dose-expansion phase | Up to 24 Moths
  ORR as measured by RECIST v1.1.

SECONDARY OUTCOMES:
PK parameters in dose-escalation phase | 240 Days
  Area Under concentration-time Curve (AUC), Maximum serum concentration (Cmax), Clearance (CL), Volume of distribution (Vd), Mean Residence Time (MRT), half-life (t1/2), time of maximum concentration (Tmax), and average plasma concentration (Cavg).
ORR assessment in dose-escalation phase | Up to 24 Months
  Overall response rate (ORR) as measured by RECIST v1.1.
DCR assessment in dose-escalation phase | Up to 24 Months
  Disease control rate (DCR) as measured by RECIST v1.1.
DOR assessment in dose-escalation phase | Up to 24 Months
  Duration of response (DOR) as measured by RECIST v1.1.
PFS assessment in dose-escalation phase | Up to 24 Months
  Progression-free survival (PFS) as measured by RECIST v1.1.
ADA assessment in dose-escalation phase | Up to 24 Months
  Anti-drug antibody (ADA) and neutralizing antibodies (Nab).
DOR assessment in dose-expansion phase | Up to 24 Months
  Duration of response (DOR) as evaluated by investigators according to RECIST v1.1
PFS assessment in dose-expansion phase | Up to 24 Months
  Progression-free survival (PFS) as evaluated by investigators according to RECIST v1.1
OS rate(12M) assessment in dose-expansion phase | 12 Months
  The 12-month OS rate (OS12m) as evaluated by investigators according to RECIST v1.1
OS assessment in dose-expansion phase | Up to 24 Months
  Overall survival (OS) as evaluated by investigators according to RECIST v1.1
ADA assessment in dose-expansion phase | 240 Days
  Anti-drug antibody (ADA) and neutralizing antibodies (Nab).
PK parameters in dose-expansion phase | 240 Days
  Area Under concentration-time Curve (AUC), Maximum serum concentration (Cmax), Clearance (CL), Volume of distribution (Vd), Mean Residence Time (MRT), half-life (t1/2)、time to maximum concentration (Tmax)、and average plasma concentration (Cavg).

CONTACTS AND LOCATIONS:
Locations (6):
- NEXT Oncology, San Antonio, Texas, United States
- China (5):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Central Hospital Affiliated to ShanDong First Medical University, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality